CLINICAL TRIAL: NCT04503863
Title: Additional Phase 1 Study of NPC-22 for High Dosage in Healthy Adult Males
Brief Title: An Additional Study of NPC-22 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NPC-22-2
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Safety and Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): Single administration of middle dose NPC-22
  Interventions: Drug: NPC-22
- Experimental 2 (Experimental): Single administration of high dose NPC-22
  Interventions: Drug: NPC-22
- Experimental 3 (Placebo Comparator): Single administration of placebo dose NPC-22
  Interventions: Drug: NPC-22 Placebo

INTERVENTIONS:
Drug: NPC-22 — Single administration of middle dose NPC-22
  Arms: Experimental 1
Drug: NPC-22 — Single administration of high dose NPC-22
  Arms: Experimental 2
Drug: NPC-22 Placebo — Single administration of NPC-22 Placebo
  Arms: Experimental 3

SUMMARY:
The purpose of this study is to examine the safety and pharmacokinetics of high dose NPC-22 administration in healthy adult males.

The effect of administration routes for pharmacokinetics will be examined in advance.

ELIGIBILITY:
Inclusion Criteria:

Japanese individuals who have been confirmed to meet all of the following criteria will be enrolled as a subject:

1. Individuals who have provided their own written informed consent
2. Individuals aged ≥20 and <40 years at the time of informed consent
3. Individuals with body weight of ≥50 kg and body mass index (BMI) (kg/m2) of ≥18.5 and <25.0
4. Individuals who were identified to have no health problem on physical examination, physical assessment, laboratory tests, or other examinations at screening by the principal investigator or a sub-investigator

Exclusion Criteria:

Japanese Individuals who meet any of the following criteria will be excluded from the study:

1. Individuals who are suffering or have a history of any skin disease or skin abnormality at the site of study drug administration (postauricular region, breast, upper arm and abdomen) that may prevent evaluation or are receiving treatment at the site of study drug administration that may prevent evaluation (e.g., topical corticosteroids)
2. Individuals who are hypersensitive to scopolamine or atropine (belladonna alkaloid) or have a complication or a history of drug allergy
3. Individuals with a complication or a history of drug abuse (use of an illicit drug) or alcohol dependence
4. Individuals with a history of severe disease that may recur during the study period
5. Individuals with any concurrent illnesses (including symptoms and findings, however excluding diseases that will not affect study evaluations such as pollinosis without manifestations and verruca)
6. Individuals who received another study drug within 180 days prior to the start of study drug administration
7. Individuals who donated blood of ≥400 mL within 12 weeks, blood of ≥200 mL within 4 weeks, or blood components within 2 weeks prior to the start of the study
8. Individuals who used any medicinal product (including over the counter drugs except for topical products) or similar product like a dietary supplement (including health food) within 7 days prior to the start of study drug administration
9. Individuals who took any food or beverage containing grapefruit or St. John's wort within 7 days prior to the start of study drug administration
10. Individuals who took any alcohol or caffeine-containing beverage within 3 days prior to the start of study drug administration
11. Individuals who smoked (used a product such as a cigarette, pipe, cigar, chewing tobacco, electronic cigarette, nicotine patch, or nicotine gum) within 90 days prior to the start of study drug administration, or do not agree to stop smoking during the study period
12. Individuals who had a positive result for HBs antigen, HCV antibody, or HIV antigen/antibody, or a positive reaction to syphilis serology or urine drug test at screening
13. Individuals who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator based on the 12-lead electrocardiogram at screening [e.g., Fridericia's corrected QT (QTcF) interval of ≥450 ms]
14. Individuals who have serum electrolyte levels (potassium, calcium, and magnesium) lower than the institutional reference values
15. Individuals who have a familial history of torsades de pointes or long QT syndrome
16. Individuals who had blood pressure, pulse rate, or body temperature at screening as specified below [1]Systolic blood pressure: <90 mmHg or ≥140 mmHg [2]Diastolic blood pressure: <40 mmHg or ≥90 mmHg [3]Pulse rate: <50 beats/min or ≥100 beats/min [4]Body temperature: <35.0°C or ≥37.1°C
17. Individuals who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator by having a deviation from the institutional reference values
18. Individuals who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator due to other reasons

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Adverse events | 0-14 days post dose
  An adverse event will refer to any unfavorable or unintended sign (including an abnormal laboratory finding and abnormality on the 12-lead ECG or in vital signs) and symptom
Body temperature | 0-14 days post dose
  Body temperature will be measured for assess the safety of single ascending dose of NPC-22
Blood pressure | 0-14 days post dose
  Blood pressure will be measured for assess the safety of single ascending dose of NPC-22
Pulse rate | 0-14 days post dose
  Pulse rate will be measured for assess the safety of single ascending dose of NPC-22
ECG | 0-14 days post dose
  RR, PR, QRS, QT and QTcF interval and heart rate will be measured for assess the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by hematology tests | 0-14 days post dose
  Hematology tests will be performed for assessment the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by blood chemistry tests | 0-14 days post dose
  Blood chemistry tests will be performed for assessment the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by urinalysis | 0-14 days post dose
  Urinalysis will be performed for assessment the safety of single ascending dose of NPC-22

SECONDARY OUTCOMES:
Observed plasma concentration | 0-14 days post dose
Observed urine concentration | 0-14 days post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Shinanokai Shinanozaka Clinic, Shinjuku-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided